CLINICAL TRIAL: NCT02133274
Title: A Phase II Randomized Controlled Trial to Evaluate a Brief Psychosocial Intervention Together With Early Palliative Care in Reducing Depressive Symptoms of Patients With Advanced Cancer Starting First Line Palliative Chemotherapy
Brief Title: A Psychosocial Intervention Plus Early Palliative Care in the Reduction of Depression of Advanced Cancer Patients
Acronym: PREPArE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned interim analysis did not show the expected benefit of intervention A over B (effect size <0.2).
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Carlos Eduardo Paiva, MD, PhD, Barretos Cancer Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GPQual-001
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Neoplasms
Keywords: Neoplasms; Early Palliative Care; Psychosocial Intervention; Symptoms; Quality of life; Depression
MeSH Terms: conditions — Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard oncologic care (No Intervention): Standard oncologic care
- Early Palliative Care (Experimental): A first medical consult at the Palliative Care Service will be scheduled after 2 to 3 weeks from the study inclusion and every 3 to 4 weeks thereafter.
  Interventions: Other: Early Palliative Care
- Psychosocial plus early Palliative Care (Experimental): Five weekly sessions of a Brief Psychosocial Intervention based of Behavioral Cognitive Therapy plus early palliative care. Regarding the early Palliative Care, a first medical consult at the Palliative Care Service will be scheduled after 2 to 3 weeks from the study inclusion and every 3 to 4 weeks thereafter.
  Interventions: Behavioral: Brief Psychosocial Intervention; Other: Early Palliative Care

INTERVENTIONS:
Behavioral: Brief Psychosocial Intervention — Five weekly sessions of a Brief Psychosocial Intervention based of Behavioral Cognitive Therapy designed specifically for the present study.
  Arms: Psychosocial plus early Palliative Care
Other: Early Palliative Care — Early integration of Palliative Care into the standard oncologic care. Patients starting first line chemotherapy will receive immediately evaluation by the board-certified palliative care physicians.
  Arms: Early Palliative Care; Psychosocial plus early Palliative Care

SUMMARY:
The purpose of this study is to determine whether a brief psychosocial intervention together with early palliative care are feasible, acceptable and effective in the reduction of depressive symptoms of patients with advanced cancers starting first line palliative chemotherapy.

DETAILED DESCRIPTION:
Patients with advanced cancer report physical, emotional, social and existential problems that may be due to the cancer itself or its treatment. Previous studies have demonstrated the benefit of early inclusion of palliative care (PC) in combination with standard oncologic care in reducing depressive symptoms, improving quality of life, increasing survival and also decreasing unnecessary invasive procedures. However, patients continue to arrive late at PC, even in large comprehensive cancer centers. One of the barriers is the stigma of PC perceived by patients and health professionals as "a place to die." The primaries objectives are to evaluate the feasibility and satisfaction of patients with advanced cancer submitted to a brief psychosocial intervention based on Cognitive Behavioral Therapy (CBT) in addition to early PC and to evaluate the impact of these interventions on the reduction of depressive symptoms. A randomized, open-label, phase II trial, with two intervention arms and a control group. It will be included 150 patients with advanced cancer initiating palliative chemotherapy who meet the selection criteria. Participants will be recruited from the outpatient oncology clinics from the Barretos Cancer Hospital and will be randomized in one of the three treatment arms: arm A, five weekly sessions of brief psychosocial interventions based on CBT in combination with early PC; arm B, early PC only; arm C, standard oncologic care. The Hospital Anxiety and Depression Scale (HADS), Patient Health Questionnaire-9 (PHQ-9), Brazilian version of the Edmonton Symptom Assessment System (ESAS-br), European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 PAL (EORTC QLQ-C15-Pal), 13-item measure of patient satisfaction (FAMCARE-P13), and the Disease Understanding Protocol, will be the instruments used for data collection. Patients will answer these instruments at baseline and after 45, 90, 120, and 180 days after randomization. An interim analysis is planned to occur after the inclusion of 20 participants with complete data in each arm; if the Cohen's effect size between the arms A and B is small (d<<0.2), the study will continue only with arms B and C.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and <75 years;
* Adequate knowledge about the cancer diagnosis;
* Starting first line palliative antineoplastic treatment;
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) ≤ 2;
* Life expectancy> 6 months and <24 months (as per the medical oncologist);
* Must have on the following diagnoses:

Metastatic or unresectable recurrent breast cancer; Stage IIIC or IV recurrent platinum-resistant ovarian cancer; Metastatic or unresectable recurrent cervix cancer; Metastatic or unresectable recurrent endometrial cancer; Metastatic or unresectable recurrent head and neck cancer (after previous radiotherapy); Hormone-refractory metastatic or unresectable recurrent prostate cancer; Metastatic or unresectable recurrent genitourinary cancer; Metastatic or unresectable recurrent non-small cell lung cancer; Extensive-stage or recurrent small cell lung cancer; Metastatic or unresectable recurrent gastrointestinal cancer;

Exclusion Criteria:

* Currently undergoing any psychological treatment due to a psychological disorder;
* Currently using antidepressants to treat depressive disorders and / or anxiety;
* Any cognitive deficit or attention problem that could interfere in the ability to answer questionnaires or understand the study aims (as per investigator);
* Current or previous established diagnosis of any of the following psychological conditions: Substance-Related Disorders; Schizophrenia and Other Psychotic Disorders; Mood Disorders (Depressive Disorders, Bipolar Disorders); Anxiety Disorders; Dissociative Disorders; Personality Disorders; and / or a history of suicide attempt;
* Patients with single resected metastasis;
* Any co-morbid condition, which, in the opinion of the investigator, could interfere with the safety, the compliance with the study or with the interpretation of the results.
* Patients unable to go to the hospital for the study visits, regardless of the reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depression symptoms on the HADS-D and PHQ-9 at day 90. | Baseline, Day 90.
Change from baseline in satisfaction with care on the FAMCARE-patient scale at days Days 45, 90, 120 and 180. | Baseline, Days 45, 90, 120 and 180.
  Evaluation of the satisfaction perceived by the patients regarding health care.
Descriptive results about feasibility of the study. | Average duration in minutes of each intervention session (both regarding Palliative Care consultation and Psychological session); number of non-attendance to the interventions (absences); reasons reported by patients for missing.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms on the HADS-D and PHQ-9 at days 45,120 and 180. | Baseline, Days 45, 120, 180.
Change from baseline in anxiety symptoms on the HADS-A at days 45,90, 120 and 180. | Baseline, Days 45, 90, 120, 180.
Proportion of patients answering that their cancer is curable as measured using an adapted instrument to evaluate Cancer Understanding. | At 90, 120 and 180 days.
  Considering that all patients included will have incurable advanced cancers, those answering that their disease is curable will be interpreted as not adequately aware of their prognosis.
Change from baseline in cancer symptoms on the ESAS at days 45,90, 120 and 180. | Baseline, Days 45, 90, 120, 180.
Change from baseline in quality of life on the EORTC QLQ-C15-Pal at days 45,90, 120 and 180. | Baseline, Days 45, 90, 120, 180.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Paiva, MD, PHD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Derived] do Carmo TM, Paiva BSR, de Oliveira CZ, Nascimento MSA, Paiva CE. The feasibility and benefit of a brief psychosocial intervention in addition to early palliative care in patients with advanced cancer to reduce depressive symptoms: a pilot randomized controlled clinical trial. BMC Cancer. 2017 Aug 23;17(1):564. doi: 10.1186/s12885-017-3560-6. PMID 28836960
- [Derived] do Carmo TM, Paiva BS, de Siqueira MR, da Rosa Lde T, de Oliveira CZ, Nascimento MS, Paiva CE. A phase II study in advanced cancer patients to evaluate the early transition to palliative care (the PREPArE trial): protocol study for a randomized controlled trial. Trials. 2015 Apr 12;16:160. doi: 10.1186/s13063-015-0655-8. PMID 25872950